CLINICAL TRIAL: NCT03955432
Title: Long-term Cardiac Monitoring in Epilepsy: Comparative Group Study to Assess Risk of Interictal and Ictal Cardiac Dysfunction
Brief Title: Long-term Cardiac Monitoring in Epilepsy
Acronym: LOOP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough recruit
Sponsor: Northwell Health (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Ruben Kuzniecky, Vice Chairperson, Neurology, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-0820
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Focal Epilepsy; Intractable Epilepsy; Epileptic Encephalopathy; Lennox Gastaut Syndrome; Symptomatic Epilepsy; Generalized Epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Drug Resistant Epilepsy; Lennox Gastaut Syndrome; Epilepsy, Generalized

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- LINQ ICM (Experimental): The LINQ ICM (Medtronic, Inc.) is a small FDA approved cardiac monitor implanted in the subcutaneous tissue of the chest wall that is designed to continuously record a single-lead ECG, monitoring the cardiac rhythm for up to three years. The device records and stores patient's rhythm on two occasions: first when programmed criteria are met and second upon patient activation. These programmable arrhythmia criteria are based on heart rate (bradycardia, tachycardia), irregularity of heart rate and duration of rate disturbance. The LINQ ICM (or future iterations) will be utilized in this study to detect arrhythmias in our study population. The LINQ ICM is approved by the FDA for use in patients where there is a suspicion of occult cardiac arrhythmias and is therefore being utilized in this study in accordance with the FDA labeling.
  Interventions: Device: Reveal LINQ ICM System

INTERVENTIONS:
Device: Reveal LINQ ICM System — The LINQ ICM (Medtronic, Inc.) is a small FDA approved cardiac monitor implanted in the subcutaneous tissue of the chest wall that is designed to continuously record a single-lead ECG, monitoring the cardiac rhythm for up to three years. The device records and stores patient's rhythm on two occasions: first when programmed criteria are met and second upon patient activation. These programmable arrhythmia criteria are based on heart rate (bradycardia, tachycardia), irregularity of heart rate and duration of rate disturbance. The LINQ ICM (or future iterations) will be utilized in this study to detect arrhythmias in our study population.

SUMMARY:
The purpose of this research study to investigate, classify, and quantify chronic cardiac rhythm disorders in three groups of patients with epilepsy (intractable focal epilepsy, controlled focal epilepsy and symptomatic generalized epilepsy). Patients with epilepsy have a higher risk for cardiac complications than the general population. With this study, we aim to understand more about these potential complications in patients with epilepsy and assess if treatments for cardiac problems should be evaluated more carefully in patients with epilepsy.

DETAILED DESCRIPTION:
Most cardiac studies have investigated patients with intractable focal epilepsy who have a high risk for co-morbidities, accidents, injury and SUDEP. This is confounded by the major antiepileptic drug burden in this population. Very little, however, is known about the risk of cardiac arrhythmias in patients with a lower seizure burden, i.e. patients with infrequent focal seizures and/or those without secondarily generalized convulsions. Furthermore, no chronic cardiac data is available in patients with epileptic encephalopathies especially given the fact that some of these patients are known to carry mutations that increase the risk for cardiac arrhythmias.In addition, periods of reduced cerebral blood flow during tachy or brady arrhythmias may exacerbate seizure severity and during. Diagnosing and treating these arrhythmias may not only prevent adverse cardiac events, but also reduce seizure burden. This study primarily aims to compare the frequency of cardiac rhythm abnormalities in patients with epilepsy of different severity, assess the long-term cardiac risk and evaluate the possible preventive role of anti-arrhythmic agents and/or cardiac pacemaker/defibrillator needs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 years with ability to consent.
2. No primary cardiac abnormality.
3. Ability to receive an implantable loop recorder and tolerate the procedure.
4. Patients with epilepsy as described by the three groups (intractable focal epilepsy, controlled focal epilepsy and symptomatic generalized epilepsy)

Exclusion Criteria:

1. Cardiac disease of any type
2. Known epilepsy genetic disorder with potential cardiac compromise
3. Major co-morbidities such as cancer, diabetes, stroke, bleeding disorder
4. Chronic psychosis
5. Severe MR without reliable caregiver monitoring (what is MR?)
6. Already included in another clinical trial that will affect the objectives of this study.
7. Life expectancy is less than 1 year

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Incidence rate of an event (i.e., arrhythmia or seizure) | During the two years of monitoring
  Ratio of the total number of observed events divided by the number of person-days at risk in that group. Arrhythmias will be classified into different categories based on the observed data. "Arrhythmia of any type", as well as specific categories of arrhythmias will be analyzed separately.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antzelevitch C, Burashnikov A. Overview of Basic Mechanisms of Cardiac Arrhythmia. Card Electrophysiol Clin. 2011 Mar 1;3(1):23-45. doi: 10.1016/j.ccep.2010.10.012. No abstract available. PMID 21892379
- [Background] Heron SE, Scheffer IE, Berkovic SF, Dibbens LM, Mulley JC. Channelopathies in idiopathic epilepsy. Neurotherapeutics. 2007 Apr;4(2):295-304. doi: 10.1016/j.nurt.2007.01.009. PMID 17395140
- [Background] Tao JX, Qian S, Baldwin M, Chen XJ, Rose S, Ebersole SH, Ebersole JS. SUDEP, suspected positional airway obstruction, and hypoventilation in postictal coma. Epilepsia. 2010 Nov;51(11):2344-7. doi: 10.1111/j.1528-1167.2010.02719.x. Epub 2010 Sep 24. PMID 21175606
- [Background] DeGiorgio CM, DeGiorgio AC. SUDEP and heart rate variability. Epilepsy Res. 2010 Aug;90(3):309-10; author reply 311-2. doi: 10.1016/j.eplepsyres.2010.03.013. Epub 2010 Apr 15. No abstract available. PMID 20399076
- [Background] So NK, Sperling MR. Ictal asystole and SUDEP. Neurology. 2007 Jul 31;69(5):423-4. doi: 10.1212/01.wnl.0000268698.04032.bc. No abstract available. PMID 17664399
- [Background] Drake ME, Reider CR, Kay A. Electrocardiography in epilepsy patients without cardiac symptoms. Seizure. 1993 Mar;2(1):63-5. doi: 10.1016/s1059-1311(05)80104-9. PMID 8162376
- [Background] Tavernor SJ, Brown SW, Tavernor RM, Gifford C. Electrocardiograph QT lengthening associated with epileptiform EEG discharges--a role in sudden unexplained death in epilepsy? Seizure. 1996 Mar;5(1):79-83. doi: 10.1016/s1059-1311(96)80067-7. PMID 8777558
- [Background] Neufeld G, Lazar JM, Chari G, Kamran H, Akajagbor E, Salciccioli L, Kassotis J, Stewart M. Cardiac repolarization indices in epilepsy patients. Cardiology. 2009;114(4):255-60. doi: 10.1159/000233236. Epub 2009 Aug 12. PMID 19672064
- [Background] Akalin F, Tirtir A, Yilmaz Y. Increased QT dispersion in epileptic children. Acta Paediatr. 2003 Aug;92(8):916-20. doi: 10.1080/08035250310003550. PMID 12948066
- [Background] Nei M, Sperling MR, Mintzer S, Ho RT. Long-term cardiac rhythm and repolarization abnormalities in refractory focal and generalized epilepsy. Epilepsia. 2012 Aug;53(8):e137-40. doi: 10.1111/j.1528-1167.2012.03561.x. Epub 2012 Jun 18. PMID 22709423
- [Background] Johnson JN, Tester DJ, Bass NE, Ackerman MJ. Cardiac channel molecular autopsy for sudden unexpected death in epilepsy. J Child Neurol. 2010 Jul;25(7):916-21. doi: 10.1177/0883073809343722. Epub 2010 Apr 15. PMID 20395638
- [Background] Velagapudi P, Turagam M, Laurence T, Kocheril A. Cardiac arrhythmias and sudden unexpected death in epilepsy (SUDEP). Pacing Clin Electrophysiol. 2012 Mar;35(3):363-70. doi: 10.1111/j.1540-8159.2011.03276.x. Epub 2011 Nov 29. PMID 22126214
- [Background] Surges R, Henneberger C, Adjei P, Scott CA, Sander JW, Walker MC. Do alterations in inter-ictal heart rate variability predict sudden unexpected death in epilepsy? Epilepsy Res. 2009 Dec;87(2-3):277-80. doi: 10.1016/j.eplepsyres.2009.08.008. Epub 2009 Sep 10. PMID 19747799
- [Background] Rugg-Gunn FJ, Simister RJ, Squirrell M, Holdright DR, Duncan JS. Cardiac arrhythmias in focal epilepsy: a prospective long-term study. Lancet. 2004 Dec 18-31;364(9452):2212-9. doi: 10.1016/S0140-6736(04)17594-6. PMID 15610808